CLINICAL TRIAL: NCT03819465
Title: A Phase IB, Open-Label, Multi-Center Study to Determine the Efficacy and Safety of Durvalumab and/or Novel Oncology Therapies, With or Without Chemotherapy, for First-Line Stage IV Non-Small Cell Lung Cancer (NSCLC) (MAGELLAN)
Brief Title: A Study of Novel Anti-cancer Agents in Patients With Previously Untreated NSCLC
Acronym: MAGELLAN
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D933IC00001; 2018-001748-74 (EudraCT Number)
Record Dates: First submitted 2018-12-13; First posted 2019-01-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Non-Small Cell Lung Cancer (NSCLC)
Keywords: First-Line Stage IV Metastatic Non-Small Cell Lung Cancer; Stage IV Metastatic Non-Small Cell Lung Cancer; Metastatic Non-Small Cell Lung Cancer; Non-Small Cell Lung Cancer; Non-Small Cell Lung; Non-Small Cell; NSCLC; Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; danvatirsen; Pemetrexed; Carboplatin; Gemcitabine; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Treatment arms for MEDI5752 (Arms A4 and B4) will enroll 42 and 60 patients, respectively. Arm B5 (AZD2936+chemotherapy) will enroll 60 patients.
  For all other treatment arms, 30 patients will be enrolled into each arm; additional patients may be enrolled in order to have 30 evaluable patients per arm (ie, dosed).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- A1 (Experimental): Durvalumab
  Interventions: Drug: Durvalumab
- A2 (Experimental): Durvalumab + danvatirsen
  Interventions: Drug: Durvalumab; Drug: Danvatirsen
- A3 (Experimental): Durvalumab + oleclumab
  Interventions: Drug: Durvalumab; Drug: Oleclumab
- A4 (Experimental): MEDI5752
  Interventions: Drug: MEDI5752
- B1 (Experimental): Durvalumab + Investigator's choice of chemotherapy
  Interventions: Drug: Durvalumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Gemcitabine; Drug: Cisplatin; Drug: Nab-paclitaxel
- B2 (Experimental): Durvalumab + Investigator's choice of chemotherapy + danvatirsen
  Interventions: Drug: Durvalumab; Drug: Danvatirsen; Drug: Pemetrexed; Drug: Carboplatin; Drug: Gemcitabine; Drug: Cisplatin; Drug: Nab-paclitaxel
- B3 (Experimental): Durvalumab + investigator's choice of chemotherapy + oleclumab
  Interventions: Drug: Durvalumab; Drug: Oleclumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Gemcitabine; Drug: Cisplatin; Drug: Nab-paclitaxel
- B4 (Experimental): MEDI5752
  Interventions: Drug: MEDI5752
- A5 (Experimental): AZD2936
  Interventions: Drug: AZD2936
- B5 (Experimental): AZD2936 + chemotherapy
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: AZD2936

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV Cohort A: Every 4 weeks (q4w) Cohort B: Every 3 weeks (q3w) for the first 4 cycles, then every 4 weeks (q4w) starting at Cycle 5 Day 1
  Other Names: MEDI4736
  Arms: A1; A2; A3; B1; B2; B3
Drug: Danvatirsen — Danvatirsen IV Loading dose Cycle 1 Day 1, Cycle 1 Day 3, and Cycle 1 Day 5 then once a week (q1w) starting at Cycle 1 Day 8
  Other Names: AZD9150
  Arms: A2; B2
Drug: Oleclumab — Oleclumab IV Cohort A: Every 2 weeks (q2w) for first 2 cycles, then every 4 weeks (q4w) starting at Cycle 3 Day 1 Cohort B: Every 3 weeks (q3w) for the first 4 cycles, then every 4 weeks (q4w) starting at Cycle 5 Day 1
  Other Names: MEDI9447
  Arms: A3; B3
Drug: MEDI5752 — MEDI5752 IV Every 3 weeks (q3w)
  Arms: A4; B4
Drug: Pemetrexed — Pemetrexed IV Day 1 of each 21-day cycle Arm B1: Day 1 of each 21-day cycle for the first 4 cycles then either every 3 weeks (q3w) or every 4 weeks (q4w) (per investigator discretion) thereafter Arm B2 and B3: Day 1 of each 21-day cycle for the first 4 cycles then Day 1 of each 28-day cycle (q4w) thereafter Arm B5: Day 1 of each 21-day cycle throughout the study
  Arms: B1; B2; B3; B5
Drug: Carboplatin — Carboplatin IV Day 1 of each 21-day cycle
  Arms: B1; B2; B3; B5
Drug: Gemcitabine — Gemcitabine IV Days 1 and 8 of each 21-day cycle
  Arms: B1; B2; B3
Drug: Cisplatin — Cisplatin IV Day 1 of each 21-day cycle
  Arms: B1; B2; B3; B5
Drug: Nab-paclitaxel — Nab-paclitaxel IV Days 1, 8, and 15 of each 21-day cycle
  Arms: B1; B2; B3
Drug: AZD2936 — AZD2936 IV
  Arms: A5; B5

SUMMARY:
This study is designed to determine the efficacy and safety of durvalumab and/or novel oncology therapies, with or without chemotherapy, for first-line Stage IV Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
This is a Phase IB, Open-Label, Multi-Center Study to Determine the Efficacy and Safety of Durvalumab and/or Novel Oncology Therapies, With or Without Chemotherapy, for First-Line Stage IV Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Stage IV NSCLC not amenable to curative surgery or radiation
* No prior chemotherapy or any other systemic therapy for metastatic NSCLC
* Prior platinum-containing adjuvant, neoadjuvant, or definitive chemoradiation for advanced disease are eligible, if progression has occurred >12 months from end of last therapy
* Known tumor PD-L1 status
* Tumors that lack activating EGFR mutations and ALK fusions or documented local test result for any other known genomic alteration for which a targeted therapy is approved in first line per local standard of care
* WHO/ECOG status at 0 or 1 at enrollment
* Life expectancy of at least 12 weeks
* Troponin I or T ≤ ULN (per institutional guidelines)

Exclusion Criteria:

* Active or prior documented autoimmune or inflammatory disorders
* History of active primary immunodeficiency
* Any prior chemotherapy or any other systemic therapy for metastatic NSCLC
* Untreated CNS metastases

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Assessment of AEs by CTCAE v5.0 | From informed consent until the safety follow-up visit 3 months after the last dose of study drug, or until the final data cut-off (DCO) date, whichever is earlier.
  Assessment of safety and tolerability of each treatment arm

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Tumor assessments every 6-9 weeks until week 48-54, then every 12 or 18 weeks, depending on treatment arm until the earliest of radiological progression, death, withdrawal of consent, or final DCO (approximately 4 months after last patient randomized).
  Assessment of the efficacy of each treatment arm according to RECIST 1.1. ORR: The percentage of evaluable patients with a confirmed Investigator-assessed visit response of CR or PR
Duration of Response (DoR) | Tumor assessments every 6-9 weeks until week 48-54, then every 12 or 18 weeks, depending on treatment arm until the earliest of radiological progression, death, withdrawal of consent, or final DCO (approximately 4 months after last patient randomized).
  Assessment of the efficacy of each treatment arm according to RECIST 1.1. DoR: Time from date of first detection of objective response until the date of objective radiological disease progression
Progression Free Survival (PFS) | Tumor assessments every 6-9 weeks until week 48-54, then every 12/18 weeks based on arm until progression, death, withdrawal or final DCO. Further PFS data will be collected until 6 months after last patient dosed or final DCO
  Assessment of the efficacy of each treatment arm according to RECIST 1.1. PFS: Time from date of treatment assignment until the date of objective radiological disease progression using RECIST 1.1 or death (by any cause in the absence of progression)
Overall Survival (OS) | OS data will be collected until death, 6 months after last patient dosed, or the final DCO date, whichever is earlier.
  OS: Time from date of treatment assignment until the date of death by any cause
Blood concentration of durvalumab and novel oncology therapies | From Cycle 1 Day 1 until Cycle 6/7 Day 1 (21-28-day cycles) depending on arm, then every 3 cycles (except for Arms A5 & B5), at end of treatment (Arms A4 & B4, A5 & B5 only), and until 3 months following treatment discontinuation, or the final DCO date.
  Drug concentration of durvalumab and novel oncology therapies
Frequency of anti-drug antibodies (ADAs) for durvalumab and applicable novel oncology therapies | From Cycle 1 Day 1 until Cycle 6/7 Day 1 (21-28-day cycles) depending on arm, then every 3 or 6 cycles (except for arms A5&B5), at end of treatment (arms A4&B4, A5&B5 only), until 3/6 months after treatment discontinuation, or the final DCO date.
  Investigation of the immunogenicity of durvalumab and each applicable novel oncology therapy in all applicable treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Patel, MD, Principal Investigator — UCSD Morres Cancer Center; Chih-Hsin Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (31):
- United States (3):
  - Research Site, Iowa City, Iowa
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
- Austria (2):
  - Research Site, Salzburg
  - Research Site, Vienna
- Research Site, Edegem, Belgium
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (3):
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (2):
  - Research Site, Cheongju-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Cho BC, Charoentum C, Kim DW, Yang CT, Dziadziuszko R, Geater SL, Mann H, Afshar-Imani B, Lyfar P, Yang JC, Patel SP. MAGELLAN arms B1 and B3: Durvalumab plus chemotherapy with and without oleclumab in treatment-naive metastatic non-small-cell lung cancer. Lung Cancer. 2026 Jan;211:108834. doi: 10.1016/j.lungcan.2025.108834. Epub 2025 Nov 7. PMID 41380462